CLINICAL TRIAL: NCT03205761
Title: A Phase II Clinical Trial to Analyse Olaparib Response in Patients With BRCA1 and/or 2 Promoter Methylation Diagnosed of Advanced Breast Cancer (COMETA-Breast Study)
Brief Title: Analysis of Olaparib Response in Patients With BRCA1 and/or 2 Promoter Methylation Diagnosed of Advanced Breast Cancer
Acronym: COMETABreast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2015-06; 2016-001407-23 (EudraCT Number); ESR-15-11274 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2017-05-09; First posted 2017-07-02 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-08

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced Breast Cancer; Triple Negative; olaparib; lynparza; BRCA; Methylation
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib (Experimental): Patients with a positive methylation status on at least one of the two genes and lacking of known deleterious or suspected deleterious mutations in both genes could be included in the study to receive olaparib tablet formulation at 600 mg total daily dose (given in two oral administrations of 300 mg every 12 hours approximately). Patients will continue to receive their treatment until objective disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent, whichever occurs first.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib tablet formulation at 600 mg total daily dose (given in two oral administrations of 300 mg every 12 hours approximately). Patients will continue to receive their treatment until objective disease progression, symptomatic deterioration, unacceptable toxicity, death or withdrawal of consent, whichever occurs first.
  Other Names: Lynparza

SUMMARY:
This is a multicenter single-arm phase II clinical trial to evaluate the efficacy and safety of olaparib in patients diagnosed of advanced triple negative breast cancer (TNBC) with methylation of BRCA1 and/or BRCA2 promoters assessed in DNA from metastatic lesions and absence of BRCA1 and 2 germline mutations.

DETAILED DESCRIPTION:
Patients must have received at least one previous regimen in the advance disease setting and must have at least one measurable lesion that can be accurately assessed according to RECIST v.1.1. Potential eligible patients will be screened to assess somatic (s) BRCA promoter methylation at an reference central laboratory. Germinal (g) BRCA mutational status will be analyzed also centrally at 'Myriad Genetics GmBh' laboratory unless the BRCA mutational status is already known based on a Myriad previous report. Patients with a positive methylation status on at least one of the two genes and lacking of known deleterious or suspected deleterious mutations in both genes could be enrolled in the study and receive olaparib.

Blood and tumor samples collected from all screened patients could be used for the biomarker analysis, including the assessment of germline methylation status and gene expression levels of BRCA1/2. An early efficacy review will be performed after 12 evaluable patients are enrolled; if at least 4 of them show tumour response, additional patients will be included to complete a total of 34 patients.

ELIGIBILITY:
Inclusion Criteria: (Any asterisked* are applicable as an inclusion criteria prior to perform the BRCA methylation testing via central testing)

1. *The patient has signed and dated the informed consent document and it has been obtained before conducting any procedure specifically for the study.
2. Female ≥ 18 years of age on day of signing informed consent.
3. Patient with histological confirmation of breast cancer with evidence of advanced disease not amenable to resection or radiation therapy with curative intent.
4. Documented Triple Negative (TN) disease by immunohistochemistry (IHC) and/or in situ hybridization based on local testing (preferably assessed on the most recent tumour biopsy available). TN is defined as negative hormone receptor status (< 1% of tumour cells with Estrogen Receptor (ER) and Progesterone Receptor (PgR) expression) and Human Epidermal growth factor Receptor 2 (HER2) negative status (defined as IHC score 0/1+ or negative by in situ hybridization defined according to local criteria).
5. Patient must have received at least one previous regimen in the advance disease setting.
6. Absence of deleterious or suspected deleterious germline mutations in BRCA1 and BRCA2. Germinal BRCA mutational status will be centrally assessed in Myriad laboratories to check eligibility unless the test has been previously performed at Myriad and absence of mutations has been determined.
7. Availability of a tumour tissue sample from the metastatic lesions (every effort should be done to obtain the sample after the previous therapeutic regimen for advanced disease) for central testing.
8. Documented methylation of BRCA1 and/or 2 promoters based on central testing by analysis on the most recent tumour from metastatic lesions available.
9. At least one lesion measurable not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) or clinical examination and which is suitable for accurate repeated measurements according to RECIST v.1.1.
10. Patient must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥ 10.0 g/dL with no blood transfusions in the past 28 days.
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase, SGOT) /Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase, SGPT) ] ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5 x ULN
    * Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:

    Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)/ serum creatinine (mg/dL) x 72; where F=0.85 for females.
11. *Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 (see protocol attachment 2)
12. *Patient must have a life expectancy ≥ 16 weeks
13. *Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

    Postmenopausal patient is defined as a woman fulfilling any one of the following criteria (based on the National Comprehensive Cancer Network (NCCN) definition of menopause 2008):
    * Prior bilateral oophorectomy.
    * Age > 60 years.
    * Age ≤ 60 years and with amenorrhea for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and follicle stimulating hormone and estradiol in the postmenopausal range.
14. Olaparib is regarded as a compound with medium/high foetal risk, patients of childbearing potential and their partners, who are sexually active, must agree to the use of 2 highly effective forms of contraception in combination as listed below. This should be started from the signing of the informed consent and continue throughout period of taking study treatment and for at least 1 month after last dose of study drug or they must totally/truly abstain from any form of sexual intercourse (see below).

    Acceptable non-hormonal birth control methods include:
    * Total sexual abstinence. Abstinence must continue for the total duration of the study treatment and for at least 1 month after one dose. Periodic abstinence (e.g., calendar ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Vasectomised sexual partner plus male condom. With participant assurance that partner received post-vasectomy confirmation of azoospermia.
    * Tubal occlusion plus male condom.
    * Intrauterine Device (IUD) plus male condom. Provided coils are copper-banded.

    Acceptable hormonal methods:
    * Normal and low dose combined oral pills plus male condom.
    * Cerazette (desogestrel) plus male condom. Cerazette is currently the only highly efficacious progesterone based pill.
    * Hormonal shot or injection (e.g., Depo-Provera) plus male condom.
    * Etonogestrel implants (e.g. Implanon or Norplan) plus male condom.
    * Norelgestromin/ethinyl estradiol (EE) transdermal system plus male condom.
    * Intrauterine system (IUS) device (e.g., levonorgestrel releasing IUS -Mirena®) plus male condom.
    * Intravaginal device plus male condom (e.g. EE and etonogestrel).
15. *Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits, laboratory tests and examinations and other study procedures including follow up.

Exclusion Criteria: (Any asterisked* are applicable as an inclusion criteria prior to perform the BRCA methylation testing via central testing)

1. Involvement in the planning and/or conduct of the study (applies to the sponsor and/or study site staff).
2. Previous enrolment in the present study.
3. Participation in another clinical study with an investigational product during the last 4 weeks.
4. *Any previous treatment with a Poly Adenosine diphosphate-Ribose Polymerase (PARP) inhibitor, including olaparib.
5. *Patients with other malignancy within the last 5 years, except: adequately treated non-melanoma skin cancer (basal cell or squamous cell carcinoma), curatively treated in-situ cancer of the cervix, ductal carcinoma in situ (DCIS), stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥ 5 years prior to study inclusion. Patients with a history of localised breast cancer with a tumor histology different to TN, with no evidence of disease for ≥ 5 years since they completed their adjuvant treatment.
6. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons), within 3 weeks prior to study treatment (or a longer period depending on the defined characteristics of the agents used).
7. Resting ECG with corrected QT interval (QTc) > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
8. *Concomitant use of known strong Cytochrome P3A (CYP3A) inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks. Please refer to section 5.5.2.1 about strong and moderate CYP3A inhibitors.
9. *Concomitant use of known strong CYP3A inducers (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents. Please refer to section 5.5.2.2 about strong and moderate CYP3A inducers.
10. *Persistent toxicities (> NCI-CTCAE grade 2) caused by previous cancer therapy (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion).
11. *Patients with myelodysplastic syndrome/acute myeloid leukaemia (MDS/AML) or with features suggestive of MDS/AML.
12. *Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Patients with brain metastases may be eligible for the study only if more than 4 weeks from treatment completion for these metastases (including radiation and/or surgery), are clinically stable at the time of study entry. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
13. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
14. *Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
15. *Breast feeding women.
16. *Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
17. *Patients with known active hepatitis (i.e., Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
18. *Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
19. *Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, moderate or severe hepatic impairment (according to Child-Pugh classification), an extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) or any psychiatric disorder that prohibits obtaining informed consent.
20. *Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
21. *Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no 10).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Complejo Hospitalario Universitario Reina Sofía
Locations (16):
- Spain (16):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario San Joan de Reus, Reus, Tarragona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Complejo Hospitalario Universitario Reina Sofía, Córdoba
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Centro Oncológico MD Anderson International España, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Zaragoza "Lozano Blesa", Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olaparib
Started | 11
Completed | 0
Not Completed | 11
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 10

BASELINE CHARACTERISTICS:
Arm/Group | Olaparib
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 51 [37 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 11
Menopause Status [Count of Participants; unit: Participants]
  Postmenopausal | 8
  Premenopausal | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death. 0. Asymptomatic
  1. Symptomatic but completely ambulatory
  2. Symptomatic, <50% in bed during the day
  3. Symptomatic, >50% in bed, but not bedbound
  4. Bedbound
  5. Death
  Participants
    ECOG 0 | 6
    ECOG 1 | 5
Histopathologic type [Count of Participants; unit: Participants]
  Ductal | 8
  Lobular | 1
  Not Available / Not Done | 1
  Adenoid Cystic Carcinoma | 1
Histologic grade [Count of Participants; unit: Participants] — Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster
  Participants
    Grade 1 | 1
    Grade 2 | 3
    Grade 3 | 7
Status at Initial Diagnosis [Count of Participants; unit: Participants]
  Without metastasis | 7
  With metastasis | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of patients with a Complete Response (CR) or Partial Response (PR) out of the patients from the efficacy population. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions.
  Tumor response will be assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1). Efficacy population is a subset of the intend to treat population that has received at least one dose of study medication and has performed at least one tumor response assessment according to RECIST v.1.1 (unless a progression, death or unacceptable toxicity is seen before the first tumor response assessment).
Time Frame: Through study treatment, and average of 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib
Number analyzed (Participants) | 11
Participants | 1

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria.
  CBR was defined as the percentage of patients with a Complete Response (CR) or Partial Response (PR) plus stable disease (SD) ≥ 24 weeks out of the efficacy population. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; SD is defined as a failure to meet criteria for CR or PR in the absence of progressive disease. Overall Response (OR) = CR + PR.
  Efficacy population is a subset of the intend to treat population that has received at least one dose of study medication and has performed at least one tumor response assessment according to RECIST v.1.1 (unless a progression, death or unacceptable toxicity is seen before the first tumor response assessment).
Time Frame: Through study treatment, and average of 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib
Number analyzed (Participants) | 11
Participants | 4

3. Secondary Outcome: Response Duration (RD)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. RD was defined as the time from the first documentation of objective tumor response (complete response (CR) or partial response (PR)) to the first documented progressive disease (PD), or to death due to any cause, whichever occurs first.
  Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; PD is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Through study treatment, up to 19 months
Population: There was only 1 Partial Response.
Measure: Number; unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 1
months | 18.4

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1). PFS is defined as the time from enrollment to the first documented progression disease (PD), or death from any cause, whichever occurs first. PD is defined using RECIST, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Through study treatment, and average of 8 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 11
months | 1.8 [1.2 to 3.7]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) defined as the time from the date of study enrollment to the date of death from any cause.
Time Frame: Up to 14 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 11
months | 8.9 [1.2 to 13.7]

6. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE) Related to Study Treatment
Description: Safety assessments were performed at baseline and during the study: blood pressure, pulse, body temperature, performance status evaluation, 12-lead electrocardiogram, hemoglobin, red blod cells, platelet, mean cell volume, mean cell haemoglobin concentration, mean cell haemoglobin, white blood cells, absolute differential white cell count, absolute neutrophil count or segmented neutrophil count and band forms, activated partial thromboplastin time, international normalised ratio, sodium, potassium, calcium, magnesium, fasting glucose, creatinine, total bilirubin, gamma glutamyltransferase, alkaline phosphatase, aspartate transaminase, alanine transaminase, urea/blood urea nitrogen, total protein, albumin and lactic dehydrogenase, urinalysis by dipstick, serum or urine pregnancy test, bone marrow or blood cytogenetic analysis.
  AEs were graded according to NCI-CTCAE (National Cancer Institute Common Terminology Criteria for AE) v. 4.03
Time Frame: Through study treatment, and average of 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib
Number analyzed (Participants) | 11
Participants | 8

7. Secondary Outcome: Correlation Value Between BRCA1 Methylation Status and Efficacy Outcome Data
Description: To evaluate the effect of methylation status with efficacy rate parameters it will be used chi-square test if both of them are quantitative, and will be used an ANOVA analysis if one variable is quantitative and the other one is qualitative.
Time Frame: Through study treatment, and average of 8 weeks
Population: Only 4 patients with Partial Response or Stable Disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib
Number analyzed (Participants) | 11
Participants
  Patients with no Response: BRCA1 methylated | 5
  Patients with no Response: BRCA1 no methylated | 2
  Patients with Partial Response or Stable: BRCA1 methylated | 4
  Patients with Partial Response or Stable: BRCA1 no methylated | 0

8. Secondary Outcome: Correlation Value Between BRCA2 Methylation Status and Efficacy Outcome Data
Description: as for outcome 7
Time Frame: Through study treatment, and average of 8 weeks
Population: Only 4 patients with Partial Response or Stable Disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib
Number analyzed (Participants) | 11
Participants
  Patients with Partial Response or Stable : BRCA2 methylated | 1
  Patients with Partial Response or Stable : BRCA2 no methylated | 3
  Patients with no Response : BRCA2 methylated | 3
  Patients with no Response : BRCA2 no methylated | 4

ADVERSE EVENTS:
Time Frame: AEs have been recorded through study treatment, an average of 8 weeks. Deaths were assessed up to 14 months.
Description: AE were reported after Informed Consent Document (ICD) and before study drugs until approximately 30 days following the discontinuation of study treatment.
Arm/Group | Olaparib
All-Cause Mortality (participants affected / at risk) | 8/11
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib (N=11)
Progression Disease (General disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Asthenia (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 2 (2)
Haemoglobin (Investigations) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (5)
Lymphoedema (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT03205761/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT03205761/SAP_001.pdf